CLINICAL TRIAL: NCT05483972
Title: Whole Prediabetes: A Precision Nutrition Approach to Test the Feasibility of Delivering a Family-Centered Whole Foods Diet in Adults With Prediabetes and Their Offspring
Brief Title: Whole Prediabetes: A Family-Centered Whole Foods Diet in Adults With Prediabetes and Their Offspring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nadia Markie Sneed, Principal Investigator, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 220475
Record Dates: First submitted 2022-07-25; First posted 2022-08-02 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole Prediabetes Diet Intervention (Experimental): The diet intervention will consist of weekly food deliveries for a total of 2-weeks. The intervention will consist of a weekly individual counseling sessions led by the team's registered dietitian nutritionist (RDN). Prior to beginning the intervention, an initial individual and/or family meeting with the RDN will be scheduled. The focus of the meeting will be for the RDN to provide information about diet instruction, meal preparation/planning, and individual and family goal setting. Meetings can occur in person, via a secure zoom videoconference, or via telephone (per participant preference) and must take place with the index parent present, as they will be responsible for taking the lead of the diet intervention or relaying the information to the primary caregiver/spouse/partner in the household who is responsible for meal preparation/cooking. Child/adolescent participants will be instructed by the RDN on how to record their dietary intake (as age-appropriate) using a food diary.
  Interventions: Behavioral: Whole Prediabetes Diet Intervention

INTERVENTIONS:
Behavioral: Whole Prediabetes Diet Intervention — Participants will be instructed by RDN on how to adhere to the diet intervention and will be provided menus and recipes. For the enrolled adults in the study, the goal is to maintain complete diet adherence during the two-week intervention. The focus for children/adolescents will be on encouragement and exposure of the diet by the index parent and any additional household parent/guardian/caregiver. Participants will receive groceries that are tailored specifically to the prescribed diet menus/recipes for each week. Foods will be distributed using either a grocery delivery service or via participant pick-up. Each household will receive enough groceries to feed a household of four-persons for each week of the intervention.

SUMMARY:
This study will address the following aims:

Aim 1: Design a family-centered whole foods diet adapted from the 2020-2025 DGA framework for 8-12 families that include an index parent (25-59 years) with medically managed prediabetes and their biological offspring (6-17 years).

Aim 2: Test the feasibility, acceptability, enrollment, retention, and completion rates of a 2-week family-centered whole foods-based diet for 8-12 families that include an index parent (25-59 years) with medically managed prediabetes and their biological offspring 6-17 years.

Aim 3: Estimate and compare differences in baseline and 2-week body mass change (e.g., BMI, BMI percentiles and Z-scores, waist circumference) and diet quality for the index parent and their enrolled biological offspring.

DETAILED DESCRIPTION:
This dietary program is based on empirical evidence showing that a diet pattern that favors minimally processed and whole foods (e.g., whole grains, fruits, vegetables, nuts) in contrast to diet patterns with greater consumption of highly refined and ultra-processed foods are attributed to greater reductions in HbA1c and fasting plasma glucose and a reduced risk for T2D. This evidence comes primarily from prospective cohort and clinical studies of 1) adult populations without diabetes (including type 2 and pre-diabetes) and 2) adult populations with active T2D. Studies of family dietary interventions for transgenerational T2D prevention are lacking.

Studies have focused primarily on structured diet patterns such as the Mediterranean style, Vegetarian or Vegan, Dietary Approaches to Stop Hypertension (DASH), carbohydrate-restricted, and low-fat. Evidence supports that the diet patterns most effective for T2D risk reduction focused on primarily whole food consumption (e.g., Mediterranean-style, Vegetarian, and DASH). Yet, less attention has been given to studying the effectiveness of the Dietary Guidelines for American's (DGA) diet pattern which forms the basis of nutrition advice in the U.S. and is the guiding nutrition framework used for federal nutrition policy. Moreover, a benefit of the recent DGA is its customizable approach to diet.

Recognizing the importance of a whole foods structured diet and the recent shift of the Dietary Guidelines for American's DGA diet pattern towards a customizable, family-centered, whole foods approach, studies that test the effectiveness of a DGA-structured diet for T2D risk reduction should be prioritized. Before conducting efficacy and effectiveness trails, pilot data is needed to determine the feasibility and acceptability of using this family-centered diet approach in a population at "high risk" for T2D. Applying a family-lens where a transgenerational approach can be used to prevent T2D is necessary.

Therefore, this program aims are to design and test the feasibility of delivering a whole foods diet pattern using a family centered approach in a population at risk for T2D- adults with prediabetes and their "at-risk" biological offspring.

ELIGIBILITY:
Inclusion Criteria:

For this study, eligible adults will be those that:

1. are 25 to 59 years of age at time of initial screen and identify as a parent to at least one (two max) biological child or adolescent 6-17 years;
2. have a body mass index of between ≥23kg/m2 to <40kg/m2;
3. have prediabetes (based on American Diabetes Association criteria of either fasting plasma glucose of ≥100 mg/dL, HgbA1c 5.7-6.4%, or 2-hour plasma glucose during 75-g oral glucose tolerance test [OGTT] 140 mg/dL to 199 mg/dL) reported within the last 6 months and confirmed by the participants medical records;
4. have no special dietary restrictions or food allergies that would prohibit consumption of a variety of foods/beverages;
5. are English speaking;
6. reside within the greater Nashville, TN area;
7. are without medical conditions that would limit participation in a diet-related study (e.g., tube feeding, dysphagia, severe food allergy causing anaphylaxis);
8. are able to participate in a two-week dietary program that requires home preparation/cooking for all meals and snacks;

For this study, eligible offspring (child(ren)/ adolescent(s)) will be those that:

1. Are 6-17 years at time of initial screen;
2. Have an index parent with prediabetes that is actively enrolled in the program;
3. have body mass index ≥5th percentile for age and gender on standardized CDC growth curves;
4. have no special dietary restrictions or food allergies that would prohibit consumption of a variety of foods/beverages;
5. have parental commitment to participate in a two-week research study;
6. are English speaking;
7. reside within the greater Nashville, TN area and live at home with their index parent during duration of 2- week study;
8. are without medical conditions that would limit participation in a diet-related study (e.g., tube feeding, dysphagia, severe food allergy causing anaphylaxis);
9. are able to participate in a two-week dietary program that includes at least dinner and snacks provided during after-school hours;

Exclusion criteria:

Adult exclusion criteria include:

1. adults outside the specified age range of <25 years or >59 years;
2. adults whose body mass index is <23kg/m2 or those with a body mass index ≥40kg/m2 as that degree of morbid obesity represents a different phenotype where dietary behavioral intervention alone may not be sufficient to achieve weight loss);
3. are not currently undergoing routine medical supervision by a licensed healthcare provider (i.e., MD, NP, PA) for a complicated diagnosis of prediabetes that requires routine glycemic monitoring or frequent healthcare visits for management/treatment;
4. adults actively participating in any type of weight loss program (dietary or physical activity) or those who participate in regular (≥120 minutes per week) moderate to vigorous physical activity (as requirements of the program include assessing weight change as a result of the diet);
5. adults with a prior history of type 2 diabetes;
6. adults who are not English speaking;
7. adults with special dietary restrictions, food allergies, or medical conditions that prohibit participation in a diet-related study;
8. adults with serious mental or neurologic illness that impairs ability to consent/participate;
9. women who are pregnant or nursing due to increased metabolic state requiring greater energy requirements;
10. adults currently taking medications to treat diabetes or to promote weight loss;
11. adults living outside the greater Nashville, TN area;
12. adults with poor visual acuity (corrected vision worse than 20/50 with Rosenbaum Screener);
13. adults who do not otherwise meet the eligibility criteria listed in sections above as determined by pre-screen;

Offspring (child[ren] and adolescent[s]) exclusion criteria include:

1. children/adolescents outside the specified age range of <6 years or >17 years;
2. children/adolescents whose body mass index is <5th percentile for age and gender on standardized CDC growth curves;
3. children/adolescents who do not have an eligible index parent participating in the study;
4. children who do not have parental commitment to participate consistently for two-weeks;
5. children/adolescents with a current or past diagnosis of diabetes mellitus (including prediabetes and type-2);
6. children/adolescents who are not English speaking;
7. children/adolescents with special dietary restrictions, food allergies, or medical conditions that prohibit participation in a diet-related study;
8. children/adolescents who display dissenting behaviors during baseline data collection;
9. children/adolescents actively participating in any type of weight loss program (medical or lifestyle);
10. children/adolescents who do not otherwise meet the eligibility criteria listed in sections above as determined by pre-screen;

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Adult and offspring adherence to the diet program | 2 weeks
  Adherence will be assessed by the number of days the National Cancer Institute's (NCI) automated self-administered 24-hour dietary recall (ASA24™) is completed to record dietary intake. The Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool is a free, web-based tool. ASA24 enables multiple, automatically coded, self-administered 24-hour diet recalls and/or single or multi-day food records, also known as food diaries.
Change in offspring diet quality pre-post intervention | Baseline to two weeks
  The Healthy Eating Index-2015 scale was calculated from collected 24-hour dietary recall data collected using the ASA24 (Automated-Self Administered Recall System) a computerized dietary assessment tool. Data was collected through Automated Self-Administered 24-hour dietary recall to calculate HEI-2015 scores. The scores range from 0 to 100, with higher scores reflecting greater adherence with dietary recommendations from the Dietary Guidelines for Americans. A score of 100 reflects high adherence and a score of 0 reflects no adherence.
Change in Adult Body Mass Index (BMI) | Baseline to two weeks
  Body mass index (BMI) is a person's weight in kilograms divided by the square of height in meters. BMI is interpreted using standard weight status categories. These categories are the same for men and women of all body types and ages. Below 18.5 : Underweight; 18.5 - 24.9: Normal or Healthy Weight; 25.0 - 29.9: Overweight; 30.0 and Above: Obese.
Change in Offspring Body Mass Index (BMI) percentiles | Baseline to two weeks
  Body mass index (BMI) is a person's weight in kilograms divided by the square of height in meters. BMI is interpreted using standard weight status categories. The CDC BMI-for-age charts for children above 2 years will be used to calculate BMI percentiles.
Change in Offspring Body Mass Index (BMI) Z Scores | Baseline to two weeks
  Body mass index (BMI) is a person's weight in kilograms divided by the square of height in meters. BMI is interpreted using standard weight status categories. The CDC BMI-for-age charts for children above 2 years will be used to calculate BMI z-scores.
Change in Adult and Offspring Waist Measurements | Baseline to two weeks
  Waist circumference will be measured in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia M Sneed, PhD, FNP-BC, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University School of Nursing, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sneed NM, Kelley R, Turner H, Piano MR, Dagostino C, Sellers A, Bonnet K, Schlundt D, Adams LE, Heerman WJ. The development and testing of a single-arm feasibility and acceptability study of a whole foods diet intervention for adults with prediabetes and their offspring. Pilot Feasibility Stud. 2024 Oct 23;10(1):130. doi: 10.1186/s40814-024-01554-9. PMID 39444044

DOCUMENTS (1):
  • Informed Consent Form (2022-07-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT05483972/ICF_000.pdf